CLINICAL TRIAL: NCT01932411
Title: Factors That Affect the Outcomes of Cardiothoracic and Vascular Surgery
Brief Title: Factors Affect Outcomes in Cardiovascular Surgery
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 483753
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; Valvular Diseases; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Identify factors that contribute to perioperative morbidity and mortality in patients undergoing cardiac surgery that involves cardiopulmonary bypass.

Identify factors that affect perioperative morbidity and mortality in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Identify factors that affect perioperative morbidity and mortality in patients undergoing cardiac surgery.

Here are some examples, but may not limited the following factors:

1. demographic data
2. perioperative medications
3. comorbidity

ELIGIBILITY:
Inclusion Criteria:

Patients greater than or equal to 18 years old that underwent cardiovascular surgery at UC Davis Medical Center from 01/01/2001 to 07/15/2013.

Patients will only be included that underwent cardiovascular surgeries with or without cardiopulmonary bypass.

Exclusion Criteria:

Patients that did not undergo cardiovascular surgeries and age< 18 years old will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing cardiovascular surgeries
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-07; Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 12 years
  in hospital, 30 day, one year and longer

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, M.D., Principal Investigator — University of California, Davis, Department of Anesthesiology and Pain Medicine
Locations (1):
- University of California Davis Health System, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/factors-that-affect-outcomes-in-cardiovascular-surgery-616013/